CLINICAL TRIAL: NCT01019421
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose Study of Lu AE58054 in Patients With Moderate Alzheimer's Disease Treated With Donepezil
Brief Title: Lu AE58054 Added to Donepezil for the Treatment for Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12936A; EudraCT 2009-011845-24 (Registry Identifier: EudraCT)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Alzheimer's Disease
Keywords: Cognition
MeSH Terms: conditions — Alzheimer Disease | interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lu AE58054 (Experimental)
  Interventions: Drug: Lu AE58054
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AE58054 — Add-on treatment to donepezil
  Arms: Lu AE58054
Drug: Placebo — Add-on treatment to donepezil
  Arms: Placebo

SUMMARY:
The purpose of this study is to accept or reject the hypothesis that Lu AE58054 improves cognition and functional outcomes in patients with moderate Alzheimer's Disease, already in treatment with donepezil.

DETAILED DESCRIPTION:
Multi-centre, randomised, double-blind, parallel-group, placebo-controlled, fixed-dose study of Lu AE58054 as add-on to donepezil. The patient has probable Alzheimer's Disease consistent with the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.

ELIGIBILITY:
Inclusion Criteria:

* The patient (or if applicable the legally acceptable representative (LAR) and if different from the responsible caregiver) and the responsible caregiver are able to read and understand the Informed Consent Form.
* The patient has a knowledgeable and reliable caregiver who will accompany the patient to all clinic visits during the study.
* The patient (or if applicable the LAR and if different from the responsible caregiver) and the responsible caregiver have signed the Informed Consent Form.
* The patient has probable AD consistent with NINCDS-ADRDA criteria.
* The patient is a man or woman, aged at least 50 years.
* The patient has been treated with donepezil on a stable dose for at least 3 months prior to screening.

Exclusion Criteria:

* The patient has evidence of any clinically significant neurodegenerative disease or other serious neurological disorders other than AD including but not limited to Lewy body dementia, fronto-temporal dementia, Parkinson's disease, Huntington's disease, major cortical stroke, major head trauma and, primary or secondary cerebral neoplasia.
* The patient has a Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) Axis I disorder other than AD including amnestic disorders, major depressive disorder, delirium, schizophrenia or schizoaffective disorder, bipolar disorder, psychosis, panic, post traumatic stress disorder or/and cognitive disorder not otherwise specified.
* The patient has clinical and radiological findings that fulfil the standards of the National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherché et l'Enseignement en Neurosciences (NINDS-AIREN) criteria for vascular dementia.
* The patient has CT or MRI evidence of hydrocephalus, stroke, a space-occupying lesion, cerebral infection or any clinically significant central nervous system disease other than AD.
* The patient has clinically significant abnormal vital signs.
* The patient has one or more laboratory values outside the normal range, based on the blood or urine samples, which are, in the investigator's judgement, considered to be clinically significant.
* The patient has a clinically significant abnormal ECG.
* The patient has an oncological diagnosis (haematological or solid tumour) that is currently being treated, or for which there has been treatment within 5 years preceding screening, or for which there is still evidence of active disease (patients with local dermatological tumours such as basal or squamous cell carcinoma may be included).
* The patient's donepezil therapy is likely to be interrupted or discontinued during the study.
* The patient has a disease or takes medication that, in the investigator's judgement, could interfere with the assessments of safety, tolerability, or efficacy.
* The patient is, in the investigator's judgement, unlikely to comply with the clinical study protocol or is unsuitable for any reason.
* The patient is a member of the site personnel or their immediate families.
* The patient is treated against his/her will (for example, by court order).
* The patient or patient caregiver is unwilling or unable to abide by the visit schedule and other requirements of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in cognition after 24 weeks | Week 24

SECONDARY OUTCOMES:
Change in global function, activities of daily living, safety and tolerability, pharmacokinetics/pharmacodynamics | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (51):
- Australia (5):
  - AU004, East Gosford
  - AU002, Heidelberg West
  - AU005, Kew
  - AU001, Nedlands
  - AU003, Woodville South
- Canada (9):
  - CA005, Toronto, Ontario
  - CA007, Burlington
  - CA006, Calgary
  - CA008, Gatineau
  - CA011, Kamloops
  - CA002, Kingston
  - CA010, Penticton
  - CA004, Sherbrooke
  - CA001, Toronto
- Czechia (8):
  - CZ001, Kladno
  - CZ002, Kutná Hora
  - CZ007, Litoměřice
  - CZ005, Prague
  - CZ008, Prague
  - CZ006, Prague
  - CZ004, Prague
  - CZ003, Rychnov nad Kněžnou
- Germany (8):
  - DE004, Ellwangen
  - DE003, Erbach im Odenwald
  - DE005, Frankfurt am Main
  - DE002, Günzburg
  - DE001, Homburg
  - DE006, Leipzig
  - DE009, Munich
  - DE007, Unterhaching
- Italy (7):
  - IT001, Brescia
  - IT005, Brescia
  - IT008, Florence
  - IT003, Genova
  - IT004, Lamezia Terme
  - IT007, Milan
  - IT002, Roma
- Poland (8):
  - PL002, Bydgoszcz
  - PL001, Krakow
  - PL007, Lublin
  - PL003, Sopot
  - PL009, Szczecin
  - PL004, Warsaw
  - PL005, Warsaw
  - PL008, Warsaw
- Spain (6):
  - ES002, Barcelona
  - ES003, Elche
  - ES004, Madrid
  - ES005, Madrid
  - ES006, Majadahonda
  - ES001, Terrassa

REFERENCES:
- [Derived] Wilkinson D, Windfeld K, Colding-Jorgensen E. Safety and efficacy of idalopirdine, a 5-HT6 receptor antagonist, in patients with moderate Alzheimer's disease (LADDER): a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2014 Nov;13(11):1092-1099. doi: 10.1016/S1474-4422(14)70198-X. Epub 2014 Oct 5. PMID 25297016